CLINICAL TRIAL: NCT06736197
Title: An Algorithmic Approach to Preoxygenation: Stepwise Addition of Pressure Support and Positive End-expiratory Pressure When Tidal Volume Breathing is Inadequate. A Randomised Controlled Trial
Brief Title: An Algorithmic Approach to Preoxygenation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Cagin Tanriverdi, Specialist, Department of Anesthesiology and Reanimation, Principal Investigator, Pamukkale University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: PamukkaleUCTanriverdi-001
Record Dates: First submitted 2024-11-14; First posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Preoxygenation; Anaesthesia Induction; Non-invasive Positive Pressure Ventilation
Keywords: anaesthesia; preoxygenation; tidal volume; PSV; PEEP

STUDY DESIGN:
Intervention Model Description: The study was performed in 200 patients planned for general anaesthesia for elective surgery, aged 18-65 years, ASA 1-2 physical status, without premedication and ETO2 <90% at the end of the 3rd minute with spontaneous TVB of 100% oxygen. The patients were randomly assigned to one of two groups (Group TVB and Group PSV) according to a computer-generated randomisation table. In the patients included in Group TVB, the tidal volume breathing was maintained for a further two minutes. Group PSV received inspiratory pressure support of 6 cm H2O for +1 min. At the end of four minutes, patients whose ETO₂ value had not reached a minimum of 90% were randomly divided once more into two groups. One group continued with PSV, while the other was administered 4 cm H₂O PEEP in addition to PSV (Group PSV+PEEP).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group TVB (Experimental): Group TVB patients who could not reach 90% ETO2 at the end of the 3rd minute were continued with tidal volume breathing.
  Interventions: Procedure: Group TVB
- Group PSV (Experimental): Group PSV received 6 cm H2O positive pressure ventilation.
  Interventions: Procedure: Group PSV
- Group PSV+PEEP (Experimental): In addition to 6 cmH2O pressure support, 4 cmH2O end-expiratory positive pressure support was added to the patients included in Group PEEP.
  Interventions: Procedure: Group PSV; Procedure: Group PSV+PEEP

INTERVENTIONS:
Procedure: Group TVB — Patients who could not reach ETO2 value 90 with tidal volume breathing for 3 min were included in Group TVB tidal volume breathing was continued for 2 min.
  Other Names: Tidal volume breathing was continued.
  Arms: Group TVB
Procedure: Group PSV — Preoxygenation was continued by providing 6cmH2O pressure support to the patients included in this group.
  Arms: Group PSV; Group PSV+PEEP
Procedure: Group PSV+PEEP — At the 4th minute, preoxygenation was continued by adding 4 cmH2O positive end-expiratory pressure to the same 6 cmH2O pressure support for 1 min in patients whose end-tidal O2 value still reached 90% and who were included in this group.
  Arms: Group PSV+PEEP

SUMMARY:
The aim of this randomized controlled trial is to evaluate an algorithmic approach to gradually adding pressure-supported ventilation and end-tidal positive pressure when conventional tidal volume breathing is insufficient for adequate preoxygenation. The main question it aims to answer is:

* Will the proportion of patients receiving preoxygenation increase?
* Will the duration of preoxygenation decrease?

Participants will;

* 200 patients who were planned to undergo general anesthesia for elective surgeries
* aged between 18 and 65 years
* ASA 1-2 physical status
* ETO2 <90% at the end of the 3rd minute with spontaneous tidal volume breathing

DETAILED DESCRIPTION:
The patients were randomly assigned to one of two groups (Group TVB and Group PSV) according to a computer-generated randomisation table. In the patients included in Group TVB, the tidal volume breathing was maintained for a further two minutes. Group PSV received inspiratory pressure support of 6 cm H2O for +1 min. At the end of four minutes, patients whose ETO₂ value had not reached a minimum of 90% were randomly divided once more into two groups. One group continued with PSV, while the other was administered 4 cm H₂O PEEP in addition to PSV (Group PSV+PEEP).

When adequate preoxygenation was achieved, the duration of preoxygenation, SpO2, end-tidal carbon dioxide (ETCO2), arterial blood pressures and heart rate values were recorded. Any adverse effects such as discomfort or gastric distension were noted.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgeries general anaesthesia was planned for a patient aged 18-65 years with ASA 1-2 physical condition.

Exclusion Criteria:

* Haemodynamically unstable, preoperative oxygen support such as increased intracranial or intraocular pressure, to be operated on by thoracic surgery have conditions in which positive pressure ventilation may be indirectly harmful, BMI≥35 kg/m2, pregnant, undergoing emergency surgery and causing leakage in mask ventilation bearded male patients were not included in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Adequate preoxygenation. | The moment when the end-tidal oxygen value of patients with insufficient preoxygenation at the end of the third minute with spontaneous tidal volume breathing is 90 and above.
  The moment of ensuring adequate preoxygenation when the end-tidal oxygen value is 90 and above.

SECONDARY OUTCOMES:
Adverse effects | Within 5 min until target preoxygenation is reached.
  Any adverse effects such as discomfort or gastric distension were noted.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
My first trial.

REFERENCES:
- [Derived] Tanriverdi C, Yuksel Tanriverdi S, Tomatir E. Preoxygenation algorithm: sequential PSV and PEEP versus tidal volume breathing. a randomized controlled trial. Perioper Med (Lond). 2025 Oct 15;14(1):111. doi: 10.1186/s13741-025-00575-z. PMID 41094613